CLINICAL TRIAL: NCT05157724
Title: Observational Study to Compare Two Prostate Laser Enucleation Techniques (Photo-vaporization of the Prostate (PLASMA) Versus HoLEP) in Terms of Overall Post-operative Urinary Incontinence
Brief Title: Observational Study to Compare Two Prostate Laser Enucleation Techniques in Terms of Urinary Incontinence
Acronym: ENUPLASMHO
Status: Withdrawn | Type: Observational
Why Stopped: organizational problems
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: ENUPLASMHO
Record Dates: First submitted 2021-11-19; First posted 2021-12-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Hyperplasia, Benign; Prostatic Adenoma
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLASMA: This technique consists of an endoscopic intervention, through the natural route (urethra).
  Interventions: Procedure: PLASMA
- HOLEP: This is a recent and difficult technique of endoscopic prostate enucleation, requiring a greater learning curve for the operators compared to PLASMA. The principle remains the same technically as the PLASMA procedure, the energy used is not electrical energy, but a laser.
  Once the adenoma has been enucleated, it can only be removed by a morcellator (additional material) which can lead to complications such as bladder perforation. This is a blade that rotates in a tube that has to cut the adenoma once it has been freed from the prostate when it is in the bladder and it can happen that this blade catches on the bladder wall and causes a bladder wound or even a perforation.

INTERVENTIONS:
Procedure: PLASMA — The aim is to remove the prostatic adenoma by enucleation, i.e. to pass through the plane between the adenoma and the prostatic capsule, as opposed to resection, which also consists of removing the adenoma, but by making small cuts in the prostatic tissue, without necessarily reaching this anatomical plane between the adenoma and the capsule. This means removing less adenoma and therefore increasing the risk of adenomatous regrowth in the long term or obtaining worse results than enucleation in the short to medium term.
  The other advantage of using this approach is that it reduces intra- and post-operative bleeding and does not require the systematic discontinuation of anti-aggregating or anticoagulant treatments prior to the operation. The field of indications is thus potentially enlarged.
  Groups: PLASMA

SUMMARY:
Benign prostatic hypertrophy or prostatic adenoma is a benign tumour that develops in the central part of the prostate. Prostatic adenoma can result in the progressive appearance of a difficulty in evacuating the bladder or frequent urges to urinate and other complications (lithiasis, haematuria, urinary retention, etc.). Surgery is indicated when medical treatment is no longer effective and in the case of complications. The endoscopic techniques for treating prostate adenoma, PLASMA and HOLEP, are recognised and recommended by the French Association of Urology and the European Association of Urology (EAU) as Gold Standard techniques in view of the good results reported in the literature, the low rate of complications compared to the other techniques, and the reduced hospitalisation rate. For prostate volumes less than 80cc, there is no difference between HOLEP and Bipolar Plasma Enucleation of the Prostate (BTUEP) in terms of International Prostate Symptom Score (IPSS), Qmax, and reoperation rate at 12 months. The surgeon's experience is the most important factor influencing the risk of complications for HOLEP. Urinary incontinence after HOLEP according to Houssin et al. is 14.5% at 3 months and 4.2% at 6 months, the risk factors identified were surgeon experience and the existence of diabetes. Comparative evaluation of the two techniques is less frequent, hence the interest of our prospective and multicentre study. In this study, the investigators hope to demonstrate a better outcome of the PLASMA technique in terms of post-operative residual urinary incontinence.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia or prostatic adenoma is a benign tumour that develops in the central part of the prostate. It usually affects men over the age of 50, with the incidence of the disease increasing with age. Prostatic adenoma may result in the progressive appearance of bladder weakness or frequent urination and other complications (lithiasis, haematuria, urine retention, etc.).

Surgery is indicated when medical treatment is no longer effective and in the case of complications.

Among the surgical interventions, several techniques are currently offered to the patient:

* transurethral monopolar resection
* transvesical adenomectomy
* HOLEP laser enucleation of the prostate
* Bipolar resection and enucleation using the Bipolar Plasma Enucleation of the Prostate (BTUEP) technique, also known as "PLASMA".

Transurethral monopolar resection is considered an obsolete technique by the learned societies, in particular because of the risk of transurethral resection of the prostate syndrom (vital risk for the patient in the event of reabsorption of the peroperative glycocoll washing liquid), the per and postoperative haemorrhagic risk, especially in patients who are on anticoagulants and/or anti-aggregants and who cannot be stopped for the prostatic procedure.

Transvesical adenomectomy has a higher bleeding risk due to the fact that it is performed in open surgery, which is much more invasive. There is a transfusion rate of 7-14%. The rate of urinary incontinence can be as high as 10% and the rate of urethral stenosis 6%.

Compared to BTUEP or HOLEP, HOLEP has a longer operating time, longer catheterisation and hospitalisation time and a higher transfusion rate for transvesical adenomectomy.

Adenomectomy should therefore only be offered if the centre has neither HOLEP nor BTUEP according to European recommendations.

The new endoscopic techniques for treating prostate adenoma, PLASMA and HOLEP, are recognised and recommended by the French Association of Urology and the European Association of Urology (EAU) as Gold Standard techniques in view of the good results reported in the literature, the low rate of complications compared with the other techniques described above, and the reduced hospitalisation rate.

For prostate volumes less than 80cc, there is no difference between HOLEP and BTUEP in terms of IPSS, Qmax, and reoperation rate at 12 months.

Compared to conventional transurethral resection of the prostate, there was a significant improvement in International Prostate Symptom Score (IPSS), quality of life (QoL), and Qmax for the BTUEP technique. These results are valid at 36, 48 and 60 months. BTUEP was also superior in terms of haemoglobin loss, duration of irrigation, duration of catheterisation and duration of hospitalisation, as well as a reduction in the post-operative retention rate and the transfusion rate. There is no greater risk of incontinence with BTUEP than with transurethral resection of the prostate.

For HOLEP, there was no significant difference in Qmax or reoperation rate compared to MTURP. Compared to BTUEP, there was no significant difference in IPSS, QOL, and Qmax according to two meta-analyses. Functional outcomes at 7 years follow-up between HOLEP and monopolar transurethral resection of the prostate (MTURP) are comparable and HOLEP has an advantage in catheterisation time, hospitalisation, loss of haemoglobin, no more urethral strictures or urge incontinence.The experience of the surgeon is the most important factor influencing the risk of complications in HOLEP.

Urinary incontinence after HOLEP according to Houssin et al. is 14.5% at 3 months and 4.2% at 6 months, the risk factors identified were surgeon experience and the existence of diabetes.

In a comparative study of HOLEP and PLASMA, 19% of incontinence was found at 3 months for HOLEP against 6% for PLASMA.

Other a study found lower rates of 5.7% for HOLEP. Based on these data, the functional outcomes of PLASMA and HOLEP are comparable. However, comparative evaluation of the two techniques is less frequent in studies which are generally retrospective or monocentric, hence the interest of our prospective and multicentric study.

By comparing two reference techniques of prostatic enucleation, HOLEP and PLASMA, the investigators hope to demonstrate in this study a better result of the PLASMA technique in terms of post-operative residual urinary incontinence. If this is demonstrated, PLASMA could overtake HOLEP, with a significantly lower material cost and a reduced learning curve.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or more and less than 80 years,
* Prostate volume 30-80 cc inclusive
* Patient who has failed medical treatment for his prostate adenoma,
* Indication for prostate enucleation (HOLEP or PLASMA)
* Patient who was informed of the study and did not object

Exclusion Criteria:

* Patient with a diagnosis of prostate cancer,
* Patient requiring monopolar or bipolar endoscopic resection,
* Patient under legal protection

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study will be allocated into 2 groups, a PLASMA arm and a HOLEP arm, depending on the technique used by each of the surgeons in the study, which depends on the technology available in the health care institution. Therefore, no randomisation is possible for this study. A balance of centres between those performing the PLASMA technique and those performing the HOLEP technique is set up (2 centres for each technology) in order to allow the inclusion of a comparable number of patients in each group.
  Recruitment will take place through the urology consultation flow or through inpatient referrals. In the latter case, patients must have been seen at least once in consultation by an investigating physician prior to the intervention to introduce them to the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall urinary incontinence (including stress urinary incontinence and urgency) between the two prostate enucleation procedures PLASMA and HOLEP at 3-month visit | At 3 months post surgery
  Pad weight testing during 3 consecutive days

SECONDARY OUTCOMES:
Overall urinary incontinence (including stress urinary incontinence and urgency) between the two prostate enucleation procedures PLASMA and HOLEP at 1 year visit | At 1 year post surgery
  Pad weight testing during 3 consecutive days
Urinary incontinence evaluated by urinary symptom profile questionnaire between the two prostate enucleation procedures PLASMA and HOLEP at 3-month visit | At 3 months post surgery
  Urinary symptom profile questionnaire
Urinary incontinence evaluated by urinary symptom profile questionnaire between the two prostate enucleation procedures PLASMA and HOLEP at 1-year visit | At 1 year post surgery
  Urinary symptom profile questionnaire
Functional evaluation evaluated by uroflowmetry between the two prostate enucleation procedures PLASMA and HOLEP at 3-month visit | At 3 months post surgery
  Uroflowmetry
Functional evaluation evaluated by uroflowmetry between the two prostate enucleation procedures PLASMA and HOLEP at 1-year visit | At 1 year post surgery
  Uroflowmetry
Functional evaluation evaluated by International Prostate Symptom Score between the two prostate enucleation procedures PLASMA and HOLEP at 3-month visit | At 3 months post surgery
  International Prostate Symptom Score
Functional evaluation evaluated by International Prostate Symptom Score between the two prostate enucleation procedures PLASMA and HOLEP at 1-year visit | At 1 year post surgery
  International Prostate Symptom Score
Intervention surgery's time between the two prostate enucleation procedures PLASMA and HOLEP | through the surgery
  Intervention time (minutes)
Hospitalisation time between the two prostate enucleation procedures PLASMA and HOLEP | through the hospital stay
  Hospitalisation time (days)
Duration of urinary catheterisation between the two prostate enucleation procedures PLASMA and HOLEP | through the surgery
  Duration of urinary catheterisation (minutes)
Quality of life evaluated by International Prostate Symptom Score between the two prostate enucleation procedures PLASMA and HOLEP at 3-month visit | At 3 months post surgery
  International Prostate Symptom Score - Quality of life dimension
Quality of life evaluated by International Prostate Symptom Score between the two prostate enucleation procedures PLASMA and HOLEP at 1-year visit | At 1 year post surgery
  International Prostate Symptom Score - Quality of life dimension
Prescription rate of anti-cholinergic treatment between the two prostate enucleation procedures PLASMA and HOLEP | through study completion, an average of 1 year
  Recording of prescriptions for anti-cholinergic treatments
Rate of re-hospitalization between the two prostate enucleation procedures PLASMA and HOLEP | through study completion, an average of 1 year
  Record of re-hospitalizations for hematuria with bladder clotting
occurrence of short-term surgical complications (within first 3 months) between the two prostate enucleation procedures PLASMA and HOLEP | Within the first 3 months
  Collection of acute urine retention, falls, bedsores, urinary tract infections, urinary incontinence
occurrence of long-term surgical complications (within first 1 year) between the two prostate enucleation procedures PLASMA and HOLEP | through study completion, an average of 1 year
  Collection of urethral stenosis
Safety evaluation between the two prostate enucleation procedures PLASMA and HOLEP | through study completion, an average of 1 year
  Record of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Soria Jérémie, MD, Principal Investigator — ELSAN Pôle Santé République - Urology
Locations (1):
- ELSAN Pôle Santé République - Urology, Clermont-Ferrand, France

REFERENCES:
- [Background] Professionals S-O. EAU Guidelines: Management of Non-neurogenic Male LUTS
- [Background] Varkarakis I, Kyriakakis Z, Delis A, Protogerou V, Deliveliotis C. Long-term results of open transvesical prostatectomy from a contemporary series of patients. Urology. 2004 Aug;64(2):306-10. doi: 10.1016/j.urology.2004.03.033. PMID 15302484
- [Background] Kuntz RM, Lehrich K, Ahyai SA. Holmium laser enucleation of the prostate versus open prostatectomy for prostates greater than 100 grams: 5-year follow-up results of a randomised clinical trial. Eur Urol. 2008 Jan;53(1):160-6. doi: 10.1016/j.eururo.2007.08.036. Epub 2007 Aug 28. PMID 17869409
- [Background] Gratzke C, Schlenker B, Seitz M, Karl A, Hermanek P, Lack N, Stief CG, Reich O. Complications and early postoperative outcome after open prostatectomy in patients with benign prostatic enlargement: results of a prospective multicenter study. J Urol. 2007 Apr;177(4):1419-22. doi: 10.1016/j.juro.2006.11.062. PMID 17382744
- [Background] Li M, Qiu J, Hou Q, Wang D, Huang W, Hu C, Li K, Gao X. Endoscopic enucleation versus open prostatectomy for treating large benign prostatic hyperplasia: a meta-analysis of randomized controlled trials. PLoS One. 2015 Mar 31;10(3):e0121265. doi: 10.1371/journal.pone.0121265. eCollection 2015. PMID 25826453
- [Background] Skolarikos A, Papachristou C, Athanasiadis G, Chalikopoulos D, Deliveliotis C, Alivizatos G. Eighteen-month results of a randomized prospective study comparing transurethral photoselective vaporization with transvesical open enucleation for prostatic adenomas greater than 80 cc. J Endourol. 2008 Oct;22(10):2333-40. doi: 10.1089/end.2008.9709. PMID 18837655
- [Background] Naspro R, Suardi N, Salonia A, Scattoni V, Guazzoni G, Colombo R, Cestari A, Briganti A, Mazzoccoli B, Rigatti P, Montorsi F. Holmium laser enucleation of the prostate versus open prostatectomy for prostates >70 g: 24-month follow-up. Eur Urol. 2006 Sep;50(3):563-8. doi: 10.1016/j.eururo.2006.04.003. Epub 2006 May 2. PMID 16713070
- [Background] Tubaro A, Carter S, Hind A, Vicentini C, Miano L. A prospective study of the safety and efficacy of suprapubic transvesical prostatectomy in patients with benign prostatic hyperplasia. J Urol. 2001 Jul;166(1):172-6. PMID 11435849
- [Background] Lin Y, Wu X, Xu A, Ren R, Zhou X, Wen Y, Zou Y, Gong M, Liu C, Su Z, Herrmann TR. Transurethral enucleation of the prostate versus transvesical open prostatectomy for large benign prostatic hyperplasia: a systematic review and meta-analysis of randomized controlled trials. World J Urol. 2016 Sep;34(9):1207-19. doi: 10.1007/s00345-015-1735-9. Epub 2015 Dec 23. PMID 26699627
- [Background] Neill MG, Gilling PJ, Kennett KM, Frampton CM, Westenberg AM, Fraundorfer MR, Wilson LC. Randomized trial comparing holmium laser enucleation of prostate with plasmakinetic enucleation of prostate for treatment of benign prostatic hyperplasia. Urology. 2006 Nov;68(5):1020-4. doi: 10.1016/j.urology.2006.06.021. Epub 2006 Nov 7. PMID 17095078
- [Background] Zhao Z, Zeng G, Zhong W, Mai Z, Zeng S, Tao X. A prospective, randomised trial comparing plasmakinetic enucleation to standard transurethral resection of the prostate for symptomatic benign prostatic hyperplasia: three-year follow-up results. Eur Urol. 2010 Nov;58(5):752-8. doi: 10.1016/j.eururo.2010.08.026. Epub 2010 Aug 20. PMID 20800340
- [Background] Li K, Wang D, Hu C, Mao Y, Li M, Si-Tu J, Huang W, Qiu W, Qiu J. A Novel Modification of Transurethral Enucleation and Resection of the Prostate in Patients With Prostate Glands Larger than 80 mL: Surgical Procedures and Clinical Outcomes. Urology. 2018 Mar;113:153-159. doi: 10.1016/j.urology.2017.11.036. Epub 2018 Jan 3. PMID 29203184
- [Background] Zhu L, Chen S, Yang S, Wu M, Ge R, Wu W, Liao L, Tan J. Electrosurgical enucleation versus bipolar transurethral resection for prostates larger than 70 ml: a prospective, randomized trial with 5-year followup. J Urol. 2013 Apr;189(4):1427-31. doi: 10.1016/j.juro.2012.10.117. Epub 2012 Oct 31. PMID 23123549
- [Background] Zhang Y, Yuan P, Ma D, Gao X, Wei C, Liu Z, Li R, Wang S, Liu J, Liu X. Efficacy and safety of enucleation vs. resection of prostate for treatment of benign prostatic hyperplasia: a meta-analysis of randomized controlled trials. Prostate Cancer Prostatic Dis. 2019 Dec;22(4):493-508. doi: 10.1038/s41391-019-0135-4. Epub 2019 Feb 28. PMID 30816336
- [Background] Tan A, Liao C, Mo Z, Cao Y. Meta-analysis of holmium laser enucleation versus transurethral resection of the prostate for symptomatic prostatic obstruction. Br J Surg. 2007 Oct;94(10):1201-8. doi: 10.1002/bjs.5916. PMID 17729384
- [Background] Qian X, Liu H, Xu D, Xu L, Huang F, He W, Qi J, Zhu Y, Xu D. Functional outcomes and complications following B-TURP versus HoLEP for the treatment of benign prostatic hyperplasia: a review of the literature and Meta-analysis. Aging Male. 2017 Sep;20(3):184-191. doi: 10.1080/13685538.2017.1295436. Epub 2017 Apr 3. PMID 28368238
- [Background] Gilling PJ, Wilson LC, King CJ, Westenberg AM, Frampton CM, Fraundorfer MR. Long-term results of a randomized trial comparing holmium laser enucleation of the prostate and transurethral resection of the prostate: results at 7 years. BJU Int. 2012 Feb;109(3):408-11. doi: 10.1111/j.1464-410X.2011.10359.x. Epub 2011 Aug 23. PMID 21883820
- [Background] Zhang X, Shen P, He Q, Yin X, Chen Z, Gui H, Shu K, Tang Q, Yang Y, Pan X, Wang J, Chen N, Zeng H. Different lasers in the treatment of benign prostatic hyperplasia: a network meta-analysis. Sci Rep. 2016 Mar 24;6:23503. doi: 10.1038/srep23503. PMID 27009501
- [Background] Yin L, Teng J, Huang CJ, Zhang X, Xu D. Holmium laser enucleation of the prostate versus transurethral resection of the prostate: a systematic review and meta-analysis of randomized controlled trials. J Endourol. 2013 May;27(5):604-11. doi: 10.1089/end.2012.0505. Epub 2013 Feb 1. PMID 23167266
- [Background] Lourenco T, Pickard R, Vale L, Grant A, Fraser C, MacLennan G, N'Dow J; Benign Prostatic Enlargement team. Alternative approaches to endoscopic ablation for benign enlargement of the prostate: systematic review of randomised controlled trials. BMJ. 2008 Jun 30;337(7660):a449. doi: 10.1136/bmj.39575.517674.BE. PMID 18595932
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Background] Elzayat EA, Elhilali MM. Holmium laser enucleation of the prostate (HoLEP): long-term results, reoperation rate, and possible impact of the learning curve. Eur Urol. 2007 Nov;52(5):1465-71. doi: 10.1016/j.eururo.2007.04.074. Epub 2007 May 4. PMID 17498867
- [Background] Du C, Jin X, Bai F, Qiu Y. Holmium laser enucleation of the prostate: the safety, efficacy, and learning experience in China. J Endourol. 2008 May;22(5):1031-6. doi: 10.1089/end.2007.0262. PMID 18377236
- [Background] Houssin V, Olivier J, Brenier M, Pierache A, Laniado M, Mouton M, Theveniaud PE, Baumert H, Mallet R, Marquette T, Villers A, Robert G, Rizk J. Predictive factors of urinary incontinence after holmium laser enucleation of the prostate: a multicentric evaluation. World J Urol. 2021 Jan;39(1):143-148. doi: 10.1007/s00345-020-03169-0. Epub 2020 Mar 26. PMID 32219512
- [Background] Patard P, Roumiguié M, Beauval JB, Sanson S, Roulette P, Teillac L, et al. Énucléation endoscopique pour hbp obstructive : comparaison holep vs plasma. Étude prospective monocentrique des résultats périopératoires et à 1 an chez 200 patients. Progrès en Urologie. 1 nov 2018;28(13):652
- [Background] Fallara G, Capogrosso P, Schifano N, Costa A, Candela L, Cazzaniga W, Boeri L, Belladelli F, Scattoni V, Salonia A, Montorsi F. Ten-year Follow-up Results After Holmium Laser Enucleation of the Prostate. Eur Urol Focus. 2021 May;7(3):612-617. doi: 10.1016/j.euf.2020.05.012. Epub 2020 Jun 21. PMID 32576532